CLINICAL TRIAL: NCT04560634
Title: Influence of Diastolic Performance on the Response to Norepinephrine for Prevention of Spinal Anesthesia-Induced Hypotension for Cesarean Delivery and Fetal Wellbeing
Brief Title: Diastolic Performance and Norepinephrine in Spinal-Induced Hypotension for Cesarean Delivery
Acronym: NORA-CS
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, SONNINO CHIARA, Registered Anesthesiologist, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 30865/19
Record Dates: First submitted 2020-09-11; First posted 2020-09-23 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Hypotension
Keywords: norepinephrine; Cesarean section; spinal anesthesia
MeSH Terms: conditions — Hypotension | interventions — Norepinephrine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Normal Diastolic Function: Diastolic Function within normal values (defined in terms of E wave and A wave velocity and Deceleration Time according to the American Society of Echocardiography and the European Association of Echocardiography)
  Interventions: Drug: Norepinephrine; Device: ClearSight®, Edwards Lifescience, Irvine, CA
- Impaired Diastolic Function: Diastolic Function with pseudonormal pattern or impaired values (defined in terms of E wave and A wave velocity and Deceleration Time according to the American Society of Echocardiography and the European Association of Echocardiography)
  Interventions: Drug: Norepinephrine; Device: ClearSight®, Edwards Lifescience, Irvine, CA

INTERVENTIONS:
Drug: Norepinephrine — Norepinephrine is administered as a continuous infusion at 0.05 mcg/kg/min and is kept to maintain systolic blood pressure within 90-120% of baseline during spinal anaesthesia. The infusion is started at the same time cerebrospinal fluid is obtained, immediately before injection of spinal medications, through a small-bore tubing connected directly to the peripheral intravenous catheter. It is stopped 5 minutes
Device: ClearSight®, Edwards Lifescience, Irvine, CA — All patients are connected to a ClearSight® monitor (ClearSight®, Edwards Lifescience, Irvine, CA) by an inflatable finger cuff placed on the midphalanx of hand middle or ring finger with no radial artery catheter and its heart reference system (HRS) is zeroed at the level of the patient's midaxillary line.
  The ClearSight® monitoring is started in the pre-anaesthesia room and calibrated for 5 minutes before recording. The monitoring continues throughout the procedure until patient transfer in the recovery room. All data are anonymously collected on a USB pen for statistical analysis.

SUMMARY:
Background and rationale: The best agent to prevent spinal-induced hypotension is still uncertain but norepinephrine showed fewer effects on heart rate and cardiac output. In septic patients norepinephrine has been shown to produce an "endogenous fluid challenge".

Objective: We aim to assess if patients with impaired diastolic function (46% of pregnant women at term) are less able to maintain indexed cardiac output in response to norepinephrine infusion during spinal-induced vasoplegia. We also aim to assess if fetal wellbeing is related to maternal cardiac output during spinal anesthesia for cesarean delivery.

Methods: We will assess by echocardiogram the diastolic function before surgery and will then start continuous non-invasive hemodynamic monitoring with a ClearSight® monitor (ClearSight®, Edwards Lifescience, Irvine, CA) and perform a fluid challenge to relate diastolic disfunction with fluid responsiveness. Hemodynamic monitoring will continue throughout the surgery. Norepinephrine infusion will start concomitantly to beginning of spinal anesthesia and will stop 5 minutes after uterotonic medication.

Outcome: We aim to assess if patients with diastolic disfunction are less able to maintain cardiac output in response to norepinephrine infusion during spinal anesthesia induced vasoplegia. We also aim to assess if fetal wellbeing is related to maternal cardiac output during spinal anesthesia for cesarean delivery.)

ELIGIBILITY:
Inclusion Criteria:

Pregnant women between the 36th and the 40th week of gestation undergoing spinal anesthesia for elective caesarian delivery.

Exclusion Criteria:

1. age < 18 yo;
2. preeclampsia;
3. eclampsia;
4. atrial fibrillation and sinus tachycardia;
5. cardiovascular diseases;
6. neuromuscular disease;
7. emergent or urgent cesarean delivery;
8. coagulopathies;
9. contraindications to spinal anesthesia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — this study only enrolls pregnant women
Study Population: All pregnant women scheduled for elective C-section at our Institution willing to participate.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Indexed Cardiac Output | Baseline/after spinal anesthesia/after delivery
  We aim to study if the diastolic performance of the heart measured by transthoracic echocardiography in healthy pregnant women at term undergoing spinal anesthesia for caesarean delivery influences the effects of norepinephrine on indexed cardiac output (CI) measured by non-invasive continuous hemodynamic monitoring.

SECONDARY OUTCOMES:
Indexed Stroke Volume | Baseline/after spinal anesthesia/after delivery
  We will correlate diastolic performance measured by transthoracic echocardiography with the response to norepinephrine of indexed stroke volume (SVI) in ml, blood pressure (BP) in mmHg and heart rate (HR) in bpm measured by non-invasive continuous hemodynamic monitoring.
Systolic Blood Pressure | Baseline/after spinal anesthesia/after delivery
  We will correlate diastolic performance measured by transthoracic echocardiography with the response to norepinephrine of blood pressure (BP) in mmHg measured by non-invasive continuous hemodynamic monitoring.
Heart Rate | Baseline/after spinal anesthesia/after delivery
  We will correlate diastolic performance measured by transthoracic echocardiography with the response to norepinephrine of heart rate (HR) in bpm measured by non-invasive continuous hemodynamic monitoring.
Apgar Scores | Decreases of Indexed Cardiac Output after spinal anesthesia
  We ought to correlate the reduction of neonatal Apgar Scores with decreases of indexed cardiac output measured by non-invasive continuous hemodynamic monitoring.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Policlinico Universitario Agostino Gemelli, Rome, Italy